CLINICAL TRIAL: NCT04511793
Title: Hepatic Artery Infusion (HAI) Program at Duke University
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled due to availability of device commercially.
Sponsor: Michael Lidsky, M.D. (Other)
Responsible Party: Sponsor-Investigator, Michael Lidsky, M.D., Assistant Professor of Surgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106190
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Colon Cancer; Liver Cancer; Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Liver Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Hepatic Artery Infusion (HAI) (Experimental): The Medtronic Synchromed II pump with the Codman® Catheter will be used to create the investigational device. The Medtronic Synchromed II pump is a surgically implantable device that allows for the delivery of high doses of chemotherapy directly to the liver, in order to treat cancer. The device is surgically implanted into a subcutaneous pocket in the abdominal wall, and the catheter is inserted into the arterial system of the liver, allowing for chemotherapeutic delivery.
  Interventions: Device: Medtronic Synchromed II pump

INTERVENTIONS:
Device: Medtronic Synchromed II pump — The pump will be placed during surgery and the pump will be filled with a combination of floxuridine (FUDR), dexamethasone, heparin, and saline.

SUMMARY:
The Duke HAI program was implemented in November 2018 and treated 30 patients in its first 17 months using the Medtronic Synchromed II device (only commercially available device suitable for HAI for cancer patients). The Duke HAI program has demonstrated safety of HAI with an overall complication rate was 19%, similar to prior published data, with all but one complication (extrahepatic perfusion) salvaged. The Investigator has also demonstrated feasibility and efficacy of a new HAI program, with 95% of patients initiating therapy with promising hepatic response and disease control rates. This protocol will enable the team to continue this program. All eligible patients will receive the synchromed II pump with a Codman catheter and chemotherapy including FUDR, dexamethasone and heparin. Systemic chemotherapy will be given per standard of care.

DETAILED DESCRIPTION:
This protocol is an interventional study for HAI therapy at Duke. The protocol is essentially for clinical treatment and the Investigator is not collecting safety and effectiveness data on the device itself. There are three primary indications for the hepatic artery infusion pump. The first are patients with unresectable, metastatic, liver-only or -dominant colorectal cancer. Although conversion to resection is a primary goal in these patients, most of these patients will die of liver disease and therefore controlling liver disease is a secondary goal to improve survival. The second group of patients are those with resectable, but high risk metastatic, liver-only or -dominant colorectal cancer. These patients are at high risk for liver recurrence, and HAI has demonstrated significant improvement in outcomes. The last group are patients with unresectable primary liver cancer, primarily intrahepatic cholangiocarcinoma. These patients have central tumors that are rarely resectable.

Eligible patients will have the following procedures performed during this study.

1. On the day of surgery, the Synchromed II pump will be implanted and the Codman® catheter placed for chemotherapy infusion.
2. During the hospital stay, patients will have:

   * Daily physical examination to evaluate for the development of complications
   * Daily blood tests to evaluate blood cell counts and liver function
   * Initiation of a proton-pump inhibitor, if not already a home medication, which will continue indefinitely
   * Assessment of side effects

Follow-Up Visits

Clinic visits and study activities will take place every 2 weeks after surgery, and include:

* Routine blood tests for blood cell counts, kidney function, and liver function
* Nuclear medicine SPECT/CT scan to confirm the pump and catheter are working properly. This is a type of scan where the images or pictures from two different types of scans are combined together.
* Start hepatic artery infusion (HAI) chemotherapy (at 2 week post-op).

HAI includes:

* Floxuridine (FUDR)
* Dexamethasone
* Heparin: (If heparin allergy, fondaparinux will be added)
* Normal saline
* Evaluation and treatment, including blood work and refilling the pump, every 2 weeks, until treatment is discontinued.

  • Systemic chemotherapy (every 2 weeks after HAI started)
* Patients with metastatic colorectal cancer will receive systemic chemotherapy that will consist of either FOLFIRI, FOLFOX, or Irinotecan/oxaliplatin.
* Patients with cholangiocarcinoma will receive Gemcitabine/Oxaliplatin or Gemcitabine alone

When the chemotherapy regimen has completed, the Synchromed II pump will be reprogrammed every 4 weeks indefinitely.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-80
* Eastern Cooperative Oncology Group score 0-1
* Fit for major surgery
* Without evidence of cirrhosis or portal hypertension
* Labs within 14 days of surgery: White blood cells ≥3 k/uL, Absolute Neutrophil Count ≥ 1.5 k/uL, Platelets ≥ 100K /uL, Creatinine ≤ 1.5 mg/dL, Total bilirubin ≤1.5 mg/dL
* Disease should be liver-only or liver-dominant
* Arterial anatomy must be suitable, determined by the surgeon
* Primary tumor may be in place in the case of colorectal liver metastases. Patients may have colorectal liver metastases (unresectable, borderline resectable, resectable), or unresectable intrahepatic cholangiocarcinoma.
* Chemotherapy completed at least 3 weeks prior to surgery.

Exclusion Criteria:

* Patients younger than 18 or older than 80 years
* Eastern Cooperative Oncology Group score 2+
* Unfit for major surgery
* Inherent liver disease with evidence of cirrhosis or portal hypertension
* Widely metastatic disease is absolutely contraindicated
* Pregnant women (Women of childbearing potential who have not completed menopause, had a hysterectomy and/or both tubes and/or both ovaries removed and have a partner who is able to father children will have a blood or urine pregnancy test performed, and it must be negative in order to continue in the study.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients Treated | Surgery to 6 months post-surgery
  Number of patients who completed HAI therapy

SECONDARY OUTCOMES:
Serious Adverse Events | Surgery to one year post-surgery
  SAEs experienced by patients receiving the synchromed II pump and HAI therapy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lidsky, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No